CLINICAL TRIAL: NCT05295849
Title: Building Habits Together: Feasibility Trial of an Integrated Mobile and Social Network Weight Loss Intervention
Brief Title: Proof-of-Concept Study of an Integrated Mobile and Social Network Weight Loss Intervention
Acronym: BHT-OWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Worcester Polytechnic Institute (Other)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H20-0060; 1R34HL145439-01A1 (NIH)
Record Dates: First submitted 2021-07-23; First posted 2022-03-25 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Obesity
Keywords: obesity; lifestyle intervention; mobile app
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: single-arm usability pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Habit App (Experimental): Habit Mobile App
  Interventions: Behavioral: Building Habits Together Online Weight Loss 6-Week Usability Trial

INTERVENTIONS:
Behavioral: Building Habits Together Online Weight Loss 6-Week Usability Trial — The intervention includes: the Facebook-delivered Diabetes Prevention Program (DPP) Lifestyle Intervention, MyFitnessPal and the Habit app. The DPP will be delivered within a counselor-led private Facebook group. It uses behavioral strategies to help participants 1) achieve a program assigned calorie goal based on amount needed to lose 1-2 pounds per week, 2) develop a healthy diet, and 3) engage in 150-300 minutes per week of moderate intensity exercise. Participants will be instructed to use MyFitnessPal for the first two weeks, the Habit app slip tracker and exercise planner for two weeks, and the Habit app problem solver for two weeks.

SUMMARY:
The purpose of this 6 week single-arm pilot is to evaluate the feasibility of the Habit app plus Facebook group intervention in 20 adults with obesity. Participants will participate in a 6-week version of the intervention which involves receiving a feed based on the Diabetes Prevention Program in a private Facebook group, access to a professional weight loss counselor in the Facebook group, MyFitnessPal, and the Habit app.

DETAILED DESCRIPTION:
The purpose of this single-arm pilot is to evaluate the feasibility of the intervention in 20 adults with obesity. We define feasibility as use of the mobile app features (dietary self-monitoring, slip tracker, and problem sharing/solving), retention, engagement (overall, problem solving), acceptability, and burden. This study will give us information that we can use to modify the intervention and our procedures before the larger pilot study. We will enroll 20 adults with obesity to participate in the 6-week pilot. Eligible participants will receive a link to complete surveys, mailed a wifi scale, and asked to provide staff with login information for the scale so weight can be recorded during assessments. They will then have a 60-minute call with a counselor to 1) download and receive training on program technology (MyFitnessPal, Habit app, and Fitbit scale) and 2) be entered into the Facebook group. Participants will participate in a 6-week version of the intervention which involves receiving a feed based on the Diabetes Prevention Program in a private Facebook group, access to a professional weight loss counselor in the Facebook group, MyFitnessPal, and the Habit app. Every Monday in the group, participants will be given one diet and one exercise goal for the week and every Sunday they will be asked to share their progress on those goals. Every Friday they will participate in a "weigh in" thread in the group. In addition to the group, for the first two weeks, participants will be asked to use MyFitnessPal; for the second two weeks, they will be asked to use the Temptation/Slip Tracker and Exercise Planner; and for the final two weeks they will be asked to use the Problem Solver. We will ask each participant to share at least one diet or exercise problem with the group over the 6 weeks and to participate in each other's problem solving posts. Participants may attend optional weekly breakout sessions where weight loss related problems will be discussed. On the final day of the intervention, a post will go up in the group asking for a volunteer who used the app enough to brainstorm how to improve it to participate in a team meeting to discuss how to improve the program. If more than one participant volunteers, one will be randomly selected to participate. After the 6-week intervention, participants will complete the weight loss problem solving skills survey, provide a final weight, and complete individual phone interviews to discuss their experience. We will convene a team meeting with the investigators, interventionists, and a participant to discuss the results and any modifications that should be made to the program before progressing to the pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old
2. BMI 30-45 kg/m2
3. has wifi connectivity at home (for wifi scale)
4. logs into Facebook at least 5 days per week over the past 2 weeks, and has posted/replied at least once a week in the past 2 weeks
5. able to participate in the study in English.

Exclusion Criteria:

1. Pregnant/lactating or plans to become pregnant during study period
2. bipolar disorder, substance abuse, psychosis, bulimia, binge eating disorder, or severe depression
3. had bariatric surgery or plans to have surgery during the study
4. currently taking medication affecting weight
5. has lost ≥10% of weight in past year
6. is participating or intends to participate in another weight loss program during the study that provides coaching or problem solving
7. chronic pain that interferes with the ability to exercise
8. Type 1 or 2 Diabetes
9. unable to make dietary changes or increase physical activity
10. unable to walk ¼ mile unaided without stopping
11. currently smokes or vapes nicotine
12. does not live in the United States
13. had major surgery in past 6 months
14. hospitalized for psychiatric reasons in past 12 months
15. has concerns about being audiotaped during the focus groups
16. does not have or not willing to create Fitbit account for study
17. unable to access smartphone at home and at work
18. does not have FB
19. has done a study with this PI before
20. has concerns about being in FB group with faculty/students of same university in which they work/attend
21. does not have smartphone
22. smartphone type/version not meeting app requirements
23. prisoner
24. unable to provide consent
25. does not complete onboarding steps for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
We will adhere to the NIH Grant Policy on Sharing of Unique Research Resources. Any unique resources will be made available immediately after publication.
  Procedures to protect the privacy of health data of individuals will be implemented to ensure NHLBI and HIPPA privacy standards are met. After the publication of outcome data, it will be made available to individuals who have IRB approval. The final dataset will be de-identified prior to sharing. Facebook participant engagement data is difficult to de-identify thus we do not intend to share it, unless we can be completely confident that participants cannot be identified.
  We will insure that data and associated documentation is available to users only under a data sharing agreement that states a commitment to: 1) using the data only for research purposes, 2) securing the data using appropriate computer protection technology; and 3) destroying the data after analyses are completed. Datasets will be stored with encryption.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately after publication
Access Criteria: After the publication of outcome data, data will be made available to individuals who have IRB approval.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Habit App
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Habit App
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Uses of the Temptation Tracker
Description: Participants were asked to use the temptation tracker on weeks 3 and 4 of the intervention. Uses were extracted from the app's backend server.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: uses of this mobile app feature
Arm/Group | Habit App
Number analyzed (Participants) | 20
uses of this mobile app feature | 9.5 (6.3)

2. Primary Outcome: Mean Number of Slips Reported
Description: Participants were asked to report whether a temptation led to a slip or if they resisted on weeks 3 and 4 of the intervention. Uses were extracted from the app's backend server.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: slips reported
Arm/Group | Habit App
Number analyzed (Participants) | 20
slips reported | 4.8 (3.5)

3. Primary Outcome: Mean Number of Temptations Resisted
Description: as for outcome 2
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: temptations resisted
Arm/Group | Habit App
Number analyzed (Participants) | 20
temptations resisted | 4.7 (6.1)

4. Primary Outcome: Mean Number of Exercises Planned
Description: Participants were asked to plan their exercise in advance on weeks 3 and 4 of the intervention. Uses were extracted from the app's backend server.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: exercises planned
Arm/Group | Habit App
Number analyzed (Participants) | 20
exercises planned | 14.0 (10.5)

5. Primary Outcome: Mean Number of Total Problems Solved
Description: Participants were asked to use the app problem solver on weeks 5 and 6 of the intervention. Uses were extracted from the app's backend server.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: problems solved
Arm/Group | Habit App
Number analyzed (Participants) | 20
problems solved | 2.9 (2)

6. Primary Outcome: Mean Number of Diet Problems Solved
Description: as for outcome 5
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: diet problems solved
Arm/Group | Habit App
Number analyzed (Participants) | 20
diet problems solved | 1.9 (1.5)

7. Primary Outcome: Mean Number of Exercise Problems Solved
Description: as for outcome 5
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: exercise problems solved
Arm/Group | Habit App
Number analyzed (Participants) | 20
exercise problems solved | 1.0 (0.5)

8. Primary Outcome: Number of Participants Saying They Agree or Strongly Agree They Would Continue to Use the Habit App if Given the Chance
Description: Participants will rate how much they agree with the statement "I would continue to use the Habit app after the study if given the chance" on 5-point Likert scales.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Habit App
Number analyzed (Participants) | 20
Participants | 11

9. Primary Outcome: Number of Participants Saying They Agree or Strongly Agree That They Would Recommend the Habit App to a Friend
Description: Participants will rate how much they agree with the following statement "I would recommend the Habit app to a friend who is trying to lose weight" on a 5-point Likert scale.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Habit App
Number analyzed (Participants) | 20
Participants | 10

10. Primary Outcome: Number of Participants Rating the Temptation and Slip Tracker as Time-consuming
Description: Participants will rate their agreement with statements about how time-consuming participation in the program and use of each component (temptation/slip tracker, problem solver, etc) is on 5-point Likert scales. This outcome counts number of participants that Strongly Agree or Agree.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Habit App
Number analyzed (Participants) | 20
Participants | 14

11. Primary Outcome: Number of Participants Rating the Problem Solver as Time-consuming
Description: Participants will rate their agreement with statements about how time-consuming participation in the program and use of each component (slip tracker, problem solver, etc) is on 5-point Likert scales. This outcome counts number of participants that Strongly Agree or Agree.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Habit App
Number analyzed (Participants) | 20
Participants | 11

12. Primary Outcome: Number of Participants Rating the Exercise Planner as Time-consuming
Description: as for outcome 11
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Habit App
Number analyzed (Participants) | 20
Participants | 11

13. Primary Outcome: Median Total Engagements in the Facebook Group
Description: Using Grytics, we will retrieve objective engagement data from the Facebook group, including the date and content of all posts, replies, reactions, and poll votes. We will calculate the total number of posts, replies, reactions, and poll votes per participant.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: total engagements
Arm/Group | Habit App
Number analyzed (Participants) | 20
total engagements | 62 [32 to 128]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Habit App
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT05295849/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT05295849/ICF_001.pdf